CLINICAL TRIAL: NCT02100124
Title: Reducing Unintended Pregnancies Through Reproductive Life Planning and Contraceptive Action Planning
Brief Title: MyNewOptions: An Online Study of Reproductive Life Planning and Contraceptive Action Planning
Acronym: MyNewOptions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Cynthia Chuang, Associate Professor of Medicine and Public Health Sciences, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CD-1304-6117; CD-1304-6117 (Other Grant/Funding Number: PCORI)
Record Dates: First submitted 2013-11-16; First posted 2014-03-31 (Estimated); Results first posted 2018-07-11 (Actual); Last update posted 2018-07-11 (Actual); Status verified 2017-09

CONDITIONS: Contraceptive Use; Unintended Pregnancy
Keywords: reproductive life planning; action planning; contraceptive use; unintended pregnancy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Reproductive Life Planning (RLP) (Experimental): RLP is an online adaptation of the Centers for Disease Control and Prevention (CDC) reproductive life planning toll that guides women to identify their reproductive goals and individual requirements for contraception.
  Interventions: Behavioral: Reproductive Life Planning (RLP); Behavioral: Contraception information
- Reproductive Life Planning Plus (RLP+) (Experimental): RLP+ additionally includes contraceptive action planning, aimed at helping women select solutions for potential problems they may encounter with contraceptive adherence.
  Interventions: Behavioral: Reproductive Life Planning (RLP); Behavioral: Contraceptive Action Planning; Behavioral: Contraception information
- Information-only control (Active Comparator): The information-only control will deliver on-line information about their contraceptive benefits coverage and information about all FDA-approved contraceptive methods.
  Interventions: Behavioral: Contraception information

INTERVENTIONS:
Behavioral: Reproductive Life Planning (RLP)
  Arms: Reproductive Life Planning (RLP); Reproductive Life Planning Plus (RLP+)
Behavioral: Contraceptive Action Planning
  Arms: Reproductive Life Planning Plus (RLP+)
Behavioral: Contraception information

SUMMARY:
The purpose of this web-based study is to determine whether reproductive life planning (RLP), with or without contraceptive action planning (RLP+), will result in reduced risk of unintended pregnancy when compared to an information-only control group.

DETAILED DESCRIPTION:
Most US families want 2 children, resulting in the average woman spending 3 decades of her life trying to avoid pregnancy. However, most women have at least one unintended pregnancy, resulting in 1.5 million abortions and 1.7 million unintended births annually. Women and couples try to avoid unintended pregnancy for a range of personal, social, and economic reasons, but also due to the increased physical and mental health effects for children that result from unintended pregnancy. Healthcare reform now requires that private health insurance companies cover all FDA-approved contraceptive methods with no copays or deductibles to the patient, creating a great opportunity for women with health insurance to get contraceptive methods they previously could not afford. In this study, women with health insurance will be randomly assigned to one of three groups: (1) Reproductive Life Planning (RLP)-women will complete a reproductive life plan that guides them to think about if and when they would want any future pregnancies, and to determine what contraceptive method(s) are best suited to them; (2) Reproductive Life Planning Plus (RLP+) which additionally includes "if-then planning," where women determine what they will do when they encounter difficult situations that make it difficult to use their contraceptive method perfectly; or (3) an information-only control group. The online format of the study allows for the potential of wide dissemination. The RLP and RLP+ interventions are expected to result in greater likelihood of contraceptive use, continuity of contraceptive use, and contraceptive adherence, and thus reduce overall risk of unintended pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* not currently pregnant
* sexually active with a male partner in the past 6 months OR anticipate being sexually active with a male partner in the next 6 months
* does not intend pregnancy in the next 12 months
* has Internet access and email address

Exclusion Criteria:

* tubal sterilization
* hysterectomy
* partner with vasectomy

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 987 (Actual)
Dates: Start 2014-04; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia H Chuang, MD, MSc, Principal Investigator — Penn State College of Medicine
Locations (1):
- Penn State College of Medicine, Hershey, Pennsylvania, United States

REFERENCES:
- [Derived] Zheng A, Nelson HN, McCall-Hosenfeld JS, Lehman EB, Chuang CH. Recent Intimate Partner Violence and Oral Contraceptive Pill Adherence in a Cohort of Reproductive-Aged Women. J Womens Health (Larchmt). 2022 Dec;31(12):1703-1709. doi: 10.1089/jwh.2021.0622. Epub 2022 Sep 20. PMID 36126298
- [Derived] Lauring JR, Lehman EB, Deimling TA, Legro RS, Chuang CH. Combined hormonal contraception use in reproductive-age women with contraindications to estrogen use. Am J Obstet Gynecol. 2016 Sep;215(3):330.e1-7. doi: 10.1016/j.ajog.2016.03.047. Epub 2016 Apr 5. PMID 27059507
- [Derived] Chuang CH, Velott DL, Weisman CS, Sciamanna CN, Legro RS, Chinchilli VM, Moos MK, Francis EB, Confer LN, Lehman EB, Armitage CJ. Reducing Unintended Pregnancies Through Web-Based Reproductive Life Planning and Contraceptive Action Planning among Privately Insured Women: Study Protocol for the MyNewOptions Randomized, Controlled Trial. Womens Health Issues. 2015 Nov-Dec;25(6):641-8. doi: 10.1016/j.whi.2015.06.010. Epub 2015 Aug 22. PMID 26307564
- [Derived] Weisman CS, Lehman EB, Legro RS, Velott DL, Chuang CH. How do pregnancy intentions affect contraceptive choices when cost is not a factor? A study of privately insured women. Contraception. 2015 Nov;92(5):501-7. doi: 10.1016/j.contraception.2015.05.007. Epub 2015 May 19. PMID 26002807

RESULTS

PARTICIPANT FLOW:
Groups:
- Reproductive Life Planning (RLP): RLP is an online adaptation of the Centers for Disease Control and Prevention (CDC) reproductive life planning toll that guides women to identify their reproductive goals and individual requirements for contraception.
  Reproductive Life Planning (RLP)
  Contraception information
- Reproductive Life Planning Plus (RLP+): RLP+ additionally includes contraceptive action planning, aimed at helping women select solutions for potential problems they may encounter with contraceptive adherence.
  Reproductive Life Planning (RLP)
  Contraceptive Action Planning
  Contraception information
- Information-only Control: The information-only control will deliver on-line information about their contraceptive benefits coverage and information about all FDA-approved contraceptive methods.
  Contraception information
Period: Overall Study
Arm/Group | Reproductive Life Planning (RLP) | Reproductive Life Planning Plus (RLP+) | Information-only Control
Started | 329 | 329 | 326
Completed | 323 | 318 | 323
Not Completed | 6 | 11 | 3
Not completed — Lost to Follow-up | 5 | 11 | 3
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Reproductive Life Planning (RLP) | Reproductive Life Planning Plus (RLP+) | Information-only Control | Total
Number analyzed (Participants) | 329 | 329 | 326 | 984
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 329 | 329 | 326 | 984
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.02 (5.95) | 27.08 (6.13) | 27.28 (5.92) | 27.13 (5.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 329 | 329 | 326 | 984
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 329 | 329 | 326 | 984

OUTCOME MEASURES:

1. Primary Outcome: Contraceptive Use
Description: Percentage of surveys with any contraceptive use
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: percentage of surveys
Arm/Group | Reproductive Life Planning (RLP) | Reproductive Life Planning Plus (RLP+) | Information-only Control
Number analyzed (Participants) | 308 | 298 | 312
percentage of surveys | 93.43 (20.59) | 94.46 (20.53) | 94.10 (19.80)
Statistical Analysis 1: Comparison: Reproductive Life Planning (RLP) vs Information-only Control; Test type: Superiority; p = 1.0, Regression, Logistic; Odds Ratio (OR) = 0.87, 95% CI 2-sided [0.56 to 1.36]
Statistical Analysis 2: Comparison: Reproductive Life Planning Plus (RLP+) vs Information-only Control; Test type: Superiority; p = 1.0, Regression, Logistic; Odds Ratio (OR) = 1.13, 95% CI 2-sided [0.70 to 1.83]
Statistical Analysis 3: Comparison: Reproductive Life Planning (RLP) vs Reproductive Life Planning Plus (RLP+); Test type: Superiority; p = 0.53, Regression, Logistic; Odds Ratio (OR) = 1.30, 95% CI 2-sided [0.82 to 2.08]

2. Secondary Outcome: Effectiveness of Contraceptive Method
Description: Percentage of surveys where most effective contraceptive method used
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: percentage of surveys
Arm/Group | Reproductive Life Planning (RLP) | Reproductive Life Planning Plus (RLP+) | Information-only Control
Number analyzed (Participants) | 308 | 298 | 312
percentage of surveys | 60.66 (45.11) | 63.93 (43.91) | 63.19 (43.22)
Statistical Analysis 1: Comparison: Reproductive Life Planning (RLP) vs Information-only Control; Test type: Superiority; p = 0.48, Regression, Logistic; Odds Ratio (OR) = 0.88, 95% CI 2-sided [0.71 to 1.09]
Statistical Analysis 2: Comparison: Reproductive Life Planning Plus (RLP+) vs Information-only Control; Test type: Superiority; p = 1.0, Regression, Logistic; Odds Ratio (OR) = 1.08, 95% CI 2-sided [0.87 to 1.35]
Statistical Analysis 3: Comparison: Reproductive Life Planning (RLP) vs Reproductive Life Planning Plus (RLP+); Test type: Superiority; p = 0.07, Regression, Logistic; Odds Ratio (OR) = 1.23, 95% CI 2-sided [0.99 to 1.53]

3. Secondary Outcome: Contraceptive Method Satisfaction
Description: percentage of surveys where very satisfied with contraceptive method
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: percentage of surveys
Arm/Group | Reproductive Life Planning (RLP) | Reproductive Life Planning Plus (RLP+) | Information-only Control
Number analyzed (Participants) | 299 | 289 | 304
percentage of surveys | 58.22 (39.39) | 57.09 (41.13) | 57.70 (39.57)
Statistical Analysis 1: Comparison: Reproductive Life Planning (RLP) vs Information-only Control; Test type: Superiority; p = 1.0, Regression, Logistic; Odds Ratio (OR) = 1.04, 95% CI 2-sided [0.84 to 1.29]
Statistical Analysis 2: Comparison: Reproductive Life Planning Plus (RLP+) vs Information-only Control; Test type: Superiority; p = 1.0, Regression, Logistic; Odds Ratio (OR) = 1.02, 95% CI 2-sided [0.82 to 1.26]
Statistical Analysis 3: Comparison: Reproductive Life Planning (RLP) vs Reproductive Life Planning Plus (RLP+); Test type: Superiority; p = 1.0, Regression, Logistic; Odds Ratio (OR) = 0.98, 95% CI 2-sided [0.79 to 1.22]

4. Secondary Outcome: Contraceptive Adherence
Description: Percentage of surveys where contraceptive adherence was high
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: percentage of surveys
Arm/Group | Reproductive Life Planning (RLP) | Reproductive Life Planning Plus (RLP+) | Information-only Control
Number analyzed (Participants) | 299 | 289 | 304
percentage of surveys | 74.02 (34.19) | 73.27 (35.54) | 76.37 (32.69)
Statistical Analysis 1: Comparison: Reproductive Life Planning (RLP) vs Information-only Control; Test type: Superiority; p = 1.0, Regression, Logistic; Odds Ratio (OR) = 1.07, 95% CI 2-sided [0.83 to 1.37]
Statistical Analysis 2: Comparison: Reproductive Life Planning Plus (RLP+) vs Information-only Control; Test type: Superiority; p = 1.0, Regression, Logistic; Odds Ratio (OR) = 1.04, 95% CI 2-sided [0.81 to 1.33]
Statistical Analysis 3: Comparison: Reproductive Life Planning (RLP) vs Reproductive Life Planning Plus (RLP+); Test type: Superiority; p = 1.0, Regression, Logistic; Odds Ratio (OR) = 0.97, 95% CI 2-sided [0.75 to 1.25]

ADVERSE EVENTS:
Time Frame: 1 year, 5 months
Arm/Group | Reproductive Life Planning (RLP) | Reproductive Life Planning Plus (RLP+) | Information-only Control
All-Cause Mortality (participants affected / at risk) | 0/329 | 0/329 | 0/326
Serious Adverse Events (participants affected / at risk) | 0/329 | 0/329 | 0/326
Other Adverse Events (participants affected / at risk) | 0/329 | 0/329 | 0/326

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No